CLINICAL TRIAL: NCT03835195
Title: Comprehensive Care in Type 1 Diabetes and Associated Outcomes: AIDDA: a Quasiexperimental Study.
Brief Title: Comprehensive Care in Type 1 Diabetes and Associated Outcomes
Acronym: AIDDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AIDDA
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Disease Management Program (Experimental): Diabetes Disease Management Program
  Interventions: Other: Diabetes Disease Management Program
- Usual Care Process (Active Comparator): Usual care process
  Interventions: Other: Usual Care Process

INTERVENTIONS:
Other: Diabetes Disease Management Program — The attention is carried out in a single physical place, in the city of Medellin. The scheme of intervention in the comprehensive Diabetes Clinic is based on the concept of disease management. The intervention is composed of 5 phases, which apply to all the patients cared for in the institution (access, reception, entry, clinical consultation, management plan, education, pharmaceutical care). The healthcare team consists of 5 endocrinologists, an endocrinologist pediatrician, 7 general practitioners trained in diabetes, 5 pharmacists trained in diabetes and certified in education for patients with diabetes and 3 nutritionists.
  Arms: Diabetes Disease Management Program
Other: Usual Care Process — The patients are treated in the cardiovascular risk clinic (general practitioners) of their Primary Healthcare Provider Institution or by specialists in internal medicine, pediatrics or endocrinology in the different Provider Institutions of Health Services of the insurance service network of health or in private doctors' offices assigned to the insurer. In some cases there is assisted consultation (general practitioner - specialist). There is no defined periodicity for follow-up; Appointments are assigned to need, according to the criteria of the treating physicians. In some cases there is remission to educational activities, not necessarily focused on type 1 diabetes.
  Arms: Usual Care Process

SUMMARY:
Quasi-experimental, retrospective, before and after study, with a control group, to evaluate the effect of an intervention based on disease management, on metabolic control and hospitalizations, in a group of patients with type Diabetes 1, attended in a Provider Institution of Health Services of the city of Medellin - Colombia.

DETAILED DESCRIPTION:
Evaluate the effect of an intervention based on the management of the disease, on metabolic control and the number of hospitalizations related to diabetes, in a group of patients with Type 1 Diabetes attended in a specialized Health Services Provider Institution in the city of Medellin - Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 1 diabetes.
* Patients affiliated to the Entity Administrator of Health Benefits Plans (EPS Sura)
* Patients with age greater than or equal to 15 years, who had been referred to the institution at the discretion of the treating physician, for poor metabolic control and had to enter a hemoglobin glycated (HbA1C) ≥ 7.0%.

Exclusion Criteria:

* Patients who at the time of recruitment were treated with continuous insulin infusion device (insulin pump) and patients with gestational diabetes were excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Differences in HbA1C value after the intervention | 4-9 months
  It was considered as a measure of the before. The last glycated hemoglobin of the patient before starting care in the health institution, when his measurement time was not more than 6 months.
  Otherwise, the value of the first HbA1C measured in the first 15 days of admission to the health institution was considered, since it reflects the level of basal glycemic control, with which the patient was referred to the institution. The post-intervention measurement corresponded to the last HbA1C measured at 4-9 months of follow-up in the institution.

SECONDARY OUTCOMES:
Proportion of patients diagnosed with dyslipidemia after the intervention | 4-9 months
  The measurement of the previous one corresponded to the diagnosis of dyslipidemia reported in the patient's clinical history before starting care in the institution. The postintervention measurement corresponded to the diagnosis of dyslipidemia reported in the clinical history at 4-9 months.
Proportion of patients with hypoglycaemia after the intervention | 4-9 months
  The measurement of the before, corresponded to the report of at least one hypoglycaemia in the patient's clinical history before starting the care in the institution. The postintervention measurement corresponded to the report of hypoglycaemia in the clinical history at 4-9 months.
  The measurement of the previous one corresponded to the diagnosis of HBP reported in the patient's clinical history before starting the care in the institution. The postintervention measurement corresponded to the diagnosis of hypertension reported in the clinical history at 4-9 months.
Number of hospitalizations associated with diabetes, after the intervention | 4-9 months
  The measurement of the before, corresponded to the number of hospitalizations associated with diabetes, in the year prior to admission to the institution. The measurement afterwards corresponded to the measurement of hospitalizations during the Clid follow-up and in the subsequent 6 months.
Proportion of patients diagnosed with hypertension after the intervention | 4-9 months
  The measurement of the previous one corresponded to the diagnosis of High Blood Pressure reported in the patient's clinical history before starting the care in the institution. The postintervention measurement corresponded to the diagnosis of hypertension reported in the clinical history at 4-9 months.
Difference in the body mass index after the intervention | 4-9 months
  The measure corresponds to the records in the admission consultation (before) and in the consultation at 4-9 months (after) in the institution.

CONTACTS AND LOCATIONS:
Overall Officials: John Jairo Zuleta Tobón, MD, Msc, Study Director — Universidad de Antioquia
Locations (1):
- Clínica Integral de Diabetes, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No